CLINICAL TRIAL: NCT06411444
Title: Effectiveness of Kidney Shaped Versus Grape Design Nasal Stents in Conjunction With Nasoalveolar Molding Appliance on Nasolabial Esthetics in Infants With Complete Unilateral Cleft Lip and Palate: A Randomized Clinical Trial
Brief Title: Effect of Different Nasal Stent Designs With Nasoalveolar Molding Appliance
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Abd El-Ghafour, Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2024-04-28; First posted 2024-05-13 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Cleft Lip; Cleft Lip and Palate
MeSH Terms: conditions — Cleft Lip

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kidney Shaped Nasal Stent (Active Comparator): Conventional NAM with kidney shaped nasal stent added to it.
  Interventions: Device: Grape Design Nasal Stent
- Grape Design Nasal Stent (Experimental): Conventional NAM with grape shaped nasal stent added to it.
  Interventions: Device: Grape Design Nasal Stent

INTERVENTIONS:
Device: Grape Design Nasal Stent — Grape Design Nasal Stent

SUMMARY:
This study is designed to compare 2 different designs of nasal stents in conjunction with nasoalveolar molding appliance regarding the changes in nose and lip esthetics in infants with cleft lip and palate.

ELIGIBILITY:
Inclusion Criteria:

* Complete unilateral cleft lip and palate.
* younger than 30 day old

Exclusion Criteria:

* Syndromic patients.
* older than 30 days old.

Ages: 0 Days to 30 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 28 (Estimated)
Dates: Start 2024-05-15 (Estimated); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
Nase and lip esthetics | Photos are planned to be taken before starting the treatment and right after finishing it.
  Measuring linear measurements on 2D photos.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided